CLINICAL TRIAL: NCT06853886
Title: Gene Discovery in CHB Patients to Identify Unknown Pathways That Lead to B and NK Cell Deregulation
Acronym: LiNKeB2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Collaborators: National Agency for Research on AIDS and Viral Hepatitis (ANRS) (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 87RI24_0023 (LiNKeB2)
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Chronic Hepatitis B Virus
Keywords: HBV; NK celles; TLR9; B cells
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HBV patient (Other): a blood sample is done during a follow-up visit
  Interventions: Other: blood sample HBV patient
- healthy volunteers (Other): a blood sample
  Interventions: Other: blood sample healthy volunteers

INTERVENTIONS:
Other: blood sample HBV patient — During a boold sample at only one follow up visit:
  * 3 tubes EDTA 10 ml per patient
  * 1 tube "Paxgene" 1ml
  * 2 dry tube per patient
  Arms: HBV patient
Other: blood sample healthy volunteers — * 3 tubes EDTA ideally age and sex matched to CHB patient.
  * 1 tube "Paxgene" 1ml
  * 2 dry tube
  Arms: healthy volunteers

SUMMARY:
Natural Killer (NK) and B cell immune responses occur during the early stages of infection and are essential to eradicate it. Yet, chronic hepatitis B (CHB) infection occurs because the antiviral immune response is insufficient. In both NK and B cell studies we will explore the genetic alterations that occur during the varied chronic stages of the disease. We believe that our findings will allow us to understand the molecular signature of NK and B cells in the context of HBV infection.

DETAILED DESCRIPTION:
Thanks to past ANRS funding we showed that both B and NK cells are dysfunctional in Hepatitis B virus (HBV) in in vitro human models and validated in patients with chronic infection. We observed that B cells responses by Toll Like Receptor 9 (TLR9) were inhibited by the HBV viral protein HBsAg. We noted the loss of TLR9 expression on all B cell subsets by HBV was mediated by loss of its promoter activity by blocking the phosphorylation of the transcription factor CREB (pCREB). Furthermore, B cell-TLR9 mediated responses such as proliferation and cytokine production were abrogated in CHB patients. For NK cells we demonstrated several significant changes in their receptor expression, loss of cytokines IFN γ, MIP1a and cytotoxicity compared to healthy donors. However, for both NK and B cell dysfunction the molecular basis and signaling pathway of this phenomenon are poorly characterized and whether this state can be reversed, a question of therapeutic importance, is unknown. We hypothesize that several molecular changes occur in NK cells from CHB patients that depend on altering the mTOR pathway by HBV and more specifically by HBsAg. Together our results from this proposal should define the genetic signatures that lead to B and NK cell function and will contribute to our understanding on immune dysfunction by HBV. In both NK and B cell studies we will explore the genetic alterations that occur during the varied chronic stages of the disease. This can only be investigated in patients including all clinical stages of CHB.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age ≥18 years old
* HBV infection or chronic HBV infection untreated or treated with a nucleoside or nucleotide analog
* Willing and able to provide written informed consent
* Affiliated with a social securityregimen

Healthy volunteer must meet all of the following inclusion criteria to be eligible for participation in this study:

* Male or female, age between 18 and 80 years
* Willing and able to provide written informed consent

Exclusion Criteria:

* Co-infection with HCV, HIV or HDV (or HBV for healthy volunteer)
* Acute hepatitis in the year preceding recruitment
* Other liver diseases : alcohol, obesity (BMI>30), diabetes, metabolic syndrome (dyslipidemia and/or known hypertension) - Underlying immunological or cancerous diseases
* Patient with a disability that prevents him/her from fully understanding the requirements of the trial - Patient under court protection, guardianship or curatorship
* Pregnant or breast-feeding women.

Secondary exclusion criteria:

* A healthy volunteer whose vaccination status does not match that expected on the basis of serological results
* Positive blood pregnancy test on inclusion
* Positive HCV, HIV or HDV test in a patient
* Positive HBV, HCV, HIV or HDV test in a healthy volunteer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
RNA sequencing of B cells from CHB patients at different stages, description of their molecular signature | At inclusion, day 0

SECONDARY OUTCOMES:
RNA sequencing of NK cells from CHB patients at different stages, description of their molecular signature (protein expression measured by flow cytometry) | At inclusion, day 0

CONTACTS AND LOCATIONS:
Overall Officials: Véronqiue LOUSTAUD-RATTI, MD, Principal Investigator — University Hospital, Limoges
Locations (3):
- France (3):
  - Centre d'Investigation Clinique, Limoges
  - Limoges University Hospital, Limoges
  - Hospice civils de Lyon, Lyon